CLINICAL TRIAL: NCT00117598
Title: An Open-Label, Randomized, Phase 3 Trial Of Intravenous Temsirolimus (CCI-779) At Two Dose Levels Compared To Investigator's Choice Therapy In Relapsed, Refractory Subjects With Mantle Cell Lymphoma (MCL)
Brief Title: Study Evaluating Temsirolimus (CCI-779) In Mantle Cell Lymphoma (MCL)
Acronym: OPTIMAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3066K1-305; NCT00326547 (obsolete NCT alias)
Record Dates: First submitted 2005-06-30; First posted 2005-07-07 (Estimated); Results first posted 2012-03-06 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Lymphoma
Keywords: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental)
  Interventions: Drug: Temsirolimus (CCI-779)
- B (Experimental)
  Interventions: Drug: Temsirolimus (CCI-779)
- C (Active Comparator)
  Interventions: Drug: Investigator's choice

INTERVENTIONS:
Drug: Temsirolimus (CCI-779) — Temsirolimus 175 mg IV once a week for 3 weeks; followed by 75 mg IV once a week
  Arms: A
Drug: Temsirolimus (CCI-779) — Temsirolimus 175 mg IV once a week for 3 weeks; followed by 25 mg IV once a week
  Arms: B
Drug: Investigator's choice — Any of the following single agent treatments:
  1. Fludarabine 25 mg/m2 IV over 30 minutes daily for 5 consecutive days, every 28 days or oral administration, as appropriate.
  2. Chlorambucil 0.1 (0.1-0.2) mg/kg PO daily for 3 to 6 weeks as required OR 0.4 (0.3 0.8) mg/kg PO every 21 to 28 days
  3. Gemcitabine 1 gm/m2 IV over 30 minutes on days 1, 8 and 15 every 28 days or day 1 and day 8 every 21 days
  4. Cyclophosphamide 300 (200-450) mg/m2 PO daily for 5 consecutive days every 21 to 28 days, OR 600 (400-1200) mg/m2 IV every 21 to 28 days
  5. Cladribine 5 mg/m2 IV daily for 5 consecutive days, every 28 days for 2-6 cycles depending on response,
  6. Etoposide 50 (50-150) mg/m2 IV daily for 3-5 days every 21 to 28 days OR 100 (50 300) mg/m2 PO daily for 3-5 days every 21 to 28 days
  7. Prednisone 40 (20-60) mg/m2 PO daily or every other day
  8. Dexamethasone 20(20-40) mg PO/IV daily for 5 consecutive days, every 14 - 28 day
  Arms: C

SUMMARY:
This is an open-label, randomized trial in relapsed refractory subjects with mantle cell lymphoma (MCL).

ELIGIBILITY:
Inclusion Criteria:

* Mantle cell lymphoma (MCL) confirmed with histology, immunophenotype, and cyclin D1 analysis
* Received 2 to 7 prior therapies which may include hematopoietic stem cell transplant (i.e. induction + consolidation + maintenance)
* Prior treatment with an alkylating agent and an anthracycline, rituximab, individually or in combination, and status that is at least one of the following:
* Primary disease refractory to at least 2 regimens;
* Refractory to at least 1 regimen after first relapse;
* Refractory or untreated after second or greater relapse;
* Refractory to first line and relapsed after second line. Chemotherapy combinations may include, but are not limited to: CHOP (Cyclophosphamide, doxorubicin, vincristine, prednisone), R-CHOP (Rituximab, Cyclophosphamide, doxorubicin, vincristine, prednisone), FCM (Fludarabine, cyclophosphamide, mitoxantrone), R-FCM (Rituximab,Fludarabine, cyclophosphamide, mitoxantrone), ICE(Ifosfamide, carboplatin, etoposide), DHAP (Dexamethasone, cisplatin, cytarabine) and hyper-CVAD (Cyclophosphamide, doxorubicin, vincristine, dexamethasone).

Exclusion Criteria:

* Subjects who are less than or equal to six month from allogeneic hematopoietic stem cell transplant and who are on immunosuppressive therapy or have evidence of graft versus host disease
* Prior investigational therapy within 3 weeks of first dose. Investigational therapy is defined as treatment that is not approved for any indication.
* Active central nervous system (CNS) metastases, as indicated by clinical symptoms, cerebral edema, requirement for corticosteroids and/or progressive growth. (Treated CNS metastases must be stable for > 2 weeks prior to Day 1.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2005-05; Primary Completion 2007-08 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (67):
- United States (19):
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Fountain Valley, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, New Milford, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Morristown, New Jersey
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Upland, Pennsylvania
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Grapevine, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Temple, Texas
  - Pfizer Investigational Site, Seattle, Washington
- Argentina (3):
  - Pfizer Investigational Site, Buenos Aires, Buenos Aires
  - Pfizer Investigational Site, Córdoba, Córdoba Province
  - Pfizer Investigational Site, Buenos Aires
- Pfizer Investigational Site, East Melbourne, Victoria, Australia
- Pfizer Investigational Site, Vienna, Austria
- Belgium (4):
  - Pfizer Investigational Site, Ghent, Belgium
  - Pfizer Investigational Site, Bruges
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Leuven
- Brazil (2):
  - Pfizer Investigational Site, Vila Buarque, São Paulo
  - Pfizer Investigational Site, Porto Alegre - RS
- Canada (7):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Greenfield Park, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
- Pfizer Investigational Site, Providencia, Santiago Metropolitan, Chile
- China (2):
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Shanghai
- France (5):
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Pierre-Bénite
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Villejuif
- Germany (3):
  - Pfizer Investigational Site, Ulm, Baden-Wurttemberg
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Mainz
- Italy (4):
  - Pfizer Investigational Site, Bologna, Italy
  - Pfizer Investigational Site, Roma, Italy
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Milan
- Pfizer Investigational Site, Rotterdam, Netherlands
- Poland (2):
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Warsaw
- Spain (5):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Pamplona, Navarre
  - Pfizer Investigational Site, Madrid
- Sweden (2):
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Uppsala
- Pfizer Investigational Site, Aarau, Switzerland
- United Kingdom (4):
  - Pfizer Investigational Site, Plymouth, Devon
  - Pfizer Investigational Site, Southampton, Hants
  - Pfizer Investigational Site, Tooting, London
  - Pfizer Investigational Site, Sutton, Surrey

REFERENCES:
- [Derived] Hess G, Coiffier B, Crump M, Gisselbrecht C, Offner F, Romaguera J, Kang L, Moran PJ. Effect of prognostic classification on temsirolimus efficacy and safety in patients with relapsed or refractory mantle cell lymphoma: a retrospective analysis. Exp Hematol Oncol. 2015 Apr 11;4:11. doi: 10.1186/s40164-015-0006-1. eCollection 2015. PMID 25938001
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3066K1-305&StudyName=Study%20Evaluating%20Temsirolimus%20%28CCI-779%29%20In%20Mantle%20Cell%20Lymphoma%20%28MCL%29

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: September 5, 2007: Sponsor conducted primary analysis of progression free survival. As a result of these preliminary data, participants receiving investigator choice therapy and those receiving 175/25 mg temsirolimus could cross over to receive treatment with 175/75 mg temsirolimus (Protocol Amendment 5).
Groups:
- Temsirolimus 175/75 mg: Temsirolimus 175 milligrams (mg) administered intravenously (IV) once weekly for 3 weeks then 75 mg temsirolimus IV once weekly until disease progression or treatment withdrawal.
- Temsirolimus 175/25 mg: Temsirolimus 175 mg IV once weekly for 3 weeks then 25 mg temsirolimus IV once weekly until disease progression or treatment withdrawal.
- Investigator's Choice: Participants received 1 single-agent treatment, chosen by investigator:
  1. Fludarabine 25 milligram per meter squared (mg/m^2) IV daily for 5 consecutive days, every 28 days or oral administration, as needed;
  2. Chlorambucil 0.1 (0.1-0.2) mg per kilogram, orally (mg/kg, PO) daily for 3 to 6 weeks as required or 0.4 (0.3-0.8) mg/kg PO every 21 to 28 days;
  3. Gemcitabine 1 g/m^2 IV on Days 1, 8, and 15, every 28 days or Days 1 and 8 every 21 days;
  4. Cyclophosphamide 300 (200-450) mg/m^2 PO daily for 5 consecutive days every 21 to 28 days, or 600 (400-1200) mg/m^2 IV every 21 to 28 days;
  5. Cladribine 5 mg/m^2 IV daily for 5 consecutive days every 28 days for 2-6 cycles;
  6. Etoposide 50 (50-150) mg/m^2 IV daily for 3-5 days every 21 to 28 days or 100 (50-300) mg/m^2 PO daily for 3-5 days every 21 to 28 days;
  7. Prednisone 40 (20-60) mg/m^2 PO daily or every other day;
  8. Dexamethasone 20 (20-40) mg PO/IV daily for 5 consecutive days every 14 to 28 days.
- Temsirolimus 175/25 mg Then 75 mg: Temsirolimus 175 mg administered IV once weekly for 3 weeks then 25 mg temsirolimus IV once weekly until treatment cross over allowed (via Protocol Amendment 5), then 75 mg temsirolimus IV once weekly until disease progression or treatment withdrawal.
- Investigator's Choice Then Temsirolimus 175/75 mg: Participants received 1 single-agent treatment chosen by investigator until treatment cross over allowed (via Protocol Amendment 5), then temsirolimus 175 mg IV once weekly for 3 weeks; then 75 mg temsirolimus IV once weekly until disease progression or treatment withdrawal.
Period: Prior to Treatment Cross Over
Arm/Group | Temsirolimus 175/75 mg | Temsirolimus 175/25 mg | Investigator's Choice | Temsirolimus 175/25 mg Then 75 mg | Investigator's Choice Then Temsirolimus 175/75 mg
Started | 57 | 56 | 56 | 0 | 0
Completed | 0 | 3 | 4 | 0 | 0
Not Completed | 57 | 53 | 52 | 0 | 0
Not completed — Death | 40 | 41 | 37 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 4 | 0 | 0
Not completed — Other | 15 | 9 | 9 | 0 | 0
Period: After Treament Cross Over
Arm/Group | Temsirolimus 175/75 mg | Temsirolimus 175/25 mg | Investigator's Choice | Temsirolimus 175/25 mg Then 75 mg | Investigator's Choice Then Temsirolimus 175/75 mg
Started | 0 | 0 | 0 | 3 | 4
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 3 | 4
Not completed — Death | 0 | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Temsirolimus 175/75 mg | Temsirolimus 175/25 mg | Investigator's Choice | Total
Number analyzed (Participants) | 57 | 56 | 56 | 169
Age, Customized [Number; unit: years]
  <65 years | 24 | 17 | 28 | 69
  >=65 years | 33 | 39 | 28 | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 8 | 32
  Male | 48 | 41 | 48 | 137

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: The period from randomization until disease progression, death or date of last contact.
Time Frame: Baseline, every 8 weeks up to Year 1, then every 12 weeks up to Year 2, and then every 6 months until tumor progression or death (up to Year 5)
Population: Intent-to-Treat (ITT) Population: All randomized participants at time of primary analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temsirolimus 175/75 mg | Temsirolimus 175/25 mg | Investigator's Choice
Number analyzed (Participants) | 54 | 54 | 54
months | 4.8 [2.9 to 7.0] | 3.7 [3.4 to 6.2] | 1.8 [1.6 to 2.0]
Statistical Analysis 1: Comparison: Temsirolimus 175/75 mg vs Investigator's Choice; Two null hypotheses (Ho) tested: 1. PFS distributions for temsirolimus 175/75 mg and investigator's choice treatment groups are identical. 2. PFS distributions for temsirolimus 175/25 mg and investigator's choice treatment groups are identical. Alternative hypothesis (Ha) for each test was that PFS distributions differed; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.25 to 0.63] — HR from a cox model adjusted for baseline stratification factors
Statistical Analysis 2: Comparison: Temsirolimus 175/25 mg vs Investigator's Choice; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.41, 95% CI 2-sided [0.26 to 0.65] — HR from a cox model adjusted for baseline stratification factors

2. Secondary Outcome: Percentage of Participants With Objective Response
Description: Assessment of complete or partial response (CR, PR) or uncomplete response (CRu) using Response Evaluation Criteria in Solid Tumors. CR: 1) No disease evident. 2) Lymph node, nodal mass regressed to normal size. 3) Previously enlarged organ ↓ size. 4) Bone marrow clear on repeat aspirate, biopsy. CRu: CR 1 and 3, at least 1 of following: Lymph node regressed >75%. Bone marrow ↑ number or aggregate size, no cytologic/architectural atypia. PR: ≥50% ↓ index lesion, no size ↑ in other nodes, liver, spleen. Splenic and hepatic nodule regressed ≥50%. No new disease.
Time Frame: as for outcome 1
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Temsirolimus 175/75 mg | Temsirolimus 175/25 mg | Investigator's Choice
Number analyzed (Participants) | 54 | 54 | 54
percentage of participants | 22.2 [11.1 to 33.3] | 5.6 [0.0 to 11.7] | 1.9 [0.0 to 5.4]
Statistical Analysis 1: Comparison: Temsirolimus 175/75 mg vs Investigator's Choice; Test type: Superiority or Other; p = 0.0019, Fisher Exact
Statistical Analysis 2: Comparison: Temsirolimus 175/25 mg vs Investigator's Choice; Test type: Superiority or Other; p = 0.6179, Fisher Exact

3. Other Pre Specified Outcome: Overall Survival (OS)
Description: Overall survival is the duration from randomization to death. For participants who are alive, overall survival is censored at the last contact.
Time Frame: Baseline up to 5 years
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temsirolimus 175/75 mg | Temsirolimus 175/25 mg | Investigator's Choice
Number analyzed (Participants) | 54 | 54 | 54
months | 11.1 [8.2 to 18.0] | 8.8 [6.4 to 14.5] | 9.5 [5.3 to 15.1]
Statistical Analysis 1: Comparison: Temsirolimus 175/75 mg vs Investigator's Choice; Test type: Superiority or Other; p = 0.3053, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.46 to 1.28] — HR from a cox model adjusted for baseline stratification factors
Statistical Analysis 2: Comparison: Temsirolimus 175/25 mg vs Investigator's Choice; Test type: Superiority or Other; p = 0.9515, Log Rank; Cox Proportional Hazard = 0.98, 95% CI 2-sided [0.60 to 1.62] — HR from a cox model adjusted for baseline stratification factors

4. Other Pre Specified Outcome: Time to Response
Description: Time between the date of randomization and the first date of objective response for participants with a confirmed objective response.
Time Frame: as for outcome 1
Population: ITT subset of participants with a confirmed objective response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temsirolimus 175/75 mg | Temsirolimus 175/25 mg | Investigator's Choice
Number analyzed (Participants) | 12 | 3 | 1
months | 3.6 [3.5 to 4.0] | 3.5 [3.5 to 4.1] | 4.0 [NA to NA] — Not Available (NA), only 1 participant with a response
Statistical Analysis 1: Comparison: Temsirolimus 175/75 mg vs Investigator's Choice; Test type: Superiority or Other; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.14 to 9.01] — HR from a cox model adjusted for baseline stratification factors
Statistical Analysis 2: Comparison: Temsirolimus 175/25 mg vs Investigator's Choice; Test type: Superiority or Other; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.10 to 13.3] — HR from a cox model adjusted for baseline stratification factors

5. Other Pre Specified Outcome: Duration of Response
Description: Time from the first documentation of objective tumor response to first date that recurrence or progressive disease (PD) was objectively documented; censored at last valid tumor assessment.
Time Frame: as for outcome 1
Population: ITT subset of participants who had a response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temsirolimus 175/75 mg | Temsirolimus 175/25 mg | Investigator's Choice
Number analyzed (Participants) | 12 | 3 | 1
months | 7.1 [4.1 to NA] — unable to calculate, data too limited for accurate assessment | 3.6 [3.2 to 10.6] | NA [NA to NA] — NA, unable to calculate, only 1 participant with a response

6. Other Pre Specified Outcome: Time to Failure (TTF)
Description: TTF is defined as the time from randomization to the date of the first documentation of Progressive Disease (PD), the date of treatment discontinuation except completion of treatment, or date of death (any cause).
Time Frame: as for outcome 1
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temsirolimus 175/75 mg | Temsirolimus 175/25 mg | Investigator's Choice
Number analyzed (Participants) | 54 | 54 | 54
months | 3.1 [2.4 to 5.5] | 3.4 [2.7 to 5.1] | 1.7 [1.4 to 1.9]
Statistical Analysis 1: Comparison: Temsirolimus 175/75 mg vs Investigator's Choice; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.23 to 0.56] — HR from a cox model adjusted for baseline stratification factors
Statistical Analysis 2: Comparison: Temsirolimus 175/25 mg vs Investigator's Choice; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.26 to 0.60] — HR from a cox model adjusted for baseline stratification factors

7. Other Pre Specified Outcome: Time to Tumor Progression (TTP)
Description: TTP: time from randomization to first documentation of objective tumor progression (including recurrence); censored at last valid tumor assessment.
Time Frame: as for outcome 1
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temsirolimus 175/75 mg | Temsirolimus 175/25 mg | Investigator's Choice
Number analyzed (Participants) | 54 | 54 | 54
months | 5.2 [4.2 to 9.1] | 3.5 [1.9 to 6.2] | 1.9 [1.6 to 2.3]
Statistical Analysis 1: Comparison: Temsirolimus 175/75 mg vs Investigator's Choice; Test type: Superiority or Other; p = 0.0004, Log Rank; Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.23 to 0.67] — HR from a cox model adjusted for baseline stratification factors
Statistical Analysis 2: Comparison: Temsirolimus 175/25 mg vs Investigator's Choice; Test type: Superiority or Other; p = 0.0712, Log Rank; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.40 to 1.04] — HR from a cox model adjusted for baseline stratification factors

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Groups:
- Temsirolimus 175/75 mg: Temsirolimus 175 milligrams (mg) administered intravenously (IV) once weekly for 3 weeks then 75 mg temsirolimus IV once weekly until disease progression or treatment withdrawal. Includes participants who received Temsirolimus 175/75 mg prior to crossover (Protocol Amendment 5).
- Temsirolimus 175/25 mg Then 75 mg: Temsirolimus 175 mg administered IV once weekly for 3 weeks then 25 mg temsirolimus IV once weekly until treatment cross over allowed (via Protocol Amendment 5), then 75 mg temsirolimus IV once weekly until disease progression or treatment withdrawal. Adverse events (AEs) presented for these participants after they crossed over to 75 mg temsirolimus IV once weekly until disease progression or treatment withdrawal.
- Investigator's Choice Then Temsirolimus 175/75 mg: Participants received 1 single-agent treatment chosen by investigator until treatment cross over allowed (via Protocol Amendment 5), then temsirolimus 175 mg IV once weekly for 3 weeks; then 75 mg temsirolimus IV once weekly until disease progression or treatment withdrawal. AEs presented for these participants after they crossed over to 75 mg temsirolimus IV once weekly until disease progression or treatment withdrawal.
Arm/Group | Temsirolimus 175/75 mg | Temsirolimus 175/25 mg | Investigator's Choice | Temsirolimus 175/25 mg Then 75 mg | Investigator's Choice Then Temsirolimus 175/75 mg
Serious Adverse Events (participants affected / at risk) | 34/57 | 34/56 | 14/54 | 1/3 | 1/4
Other Adverse Events (participants affected / at risk) | 57/57 | 56/56 | 52/54 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temsirolimus 175/75 mg (N=57) | Temsirolimus 175/25 mg (N=56) | Investigator's Choice (N=54) | Temsirolimus 175/25 mg Then 75 mg (N=3) | Investigator's Choice Then Temsirolimus 175/75 mg (N=4)
Abdominal Pain (General disorders) | 1 | 0 | 0 | 0 | 0 — Body as a whole
Accidental Injury (General disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 3 | 2 | 0 | 0
Back Pain (General disorders) | 0 | 2 | 0 | 0 | 0
Cellulitis (General disorders) | 2 | 0 | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 1 | 0 | 0
Fever (General disorders) | 8 | 7 | 1 | 0 | 0
General Physical Health Deterioration (General disorders) | 3 | 3 | 1 | 0 | 0
Headache (General disorders) | 1 | 0 | 0 | 0 | 0
Infection (General disorders) | 3 | 2 | 2 | 0 | 1
Neutropenic Fever (General disorders) | 3 | 1 | 1 | 0 | 0
Sepsis (General disorders) | 2 | 1 | 1 | 0 | 0
Septic Shock (General disorders) | 1 | 1 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 — Cardiovascular System
Atrial Flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cerebrovascular Accident (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Endocarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Heart Failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Hypervolemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary Embolus (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Anorexia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 — Digestive System
Diarrhea (Gastrointestinal disorders) | 4 | 4 | 0 | 0 | 0
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Liver Function Tests Abnormal (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Melena (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rectal Disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ulcerative Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Acute Lymphoblastic Leukemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 — Hemic And Lymphatic System
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Lymphoma (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 0 | 0
Creatinine Increased (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 — Metabolic And Nutritional
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Edema (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0
Peripheral Edema (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Facial Paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 — Nervous System
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 — Respiratory System
Carcinoma Of Lung (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Cough Increased (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Eosinophilic Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Interstitial Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Lung Edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Lung Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Lung Infiltration Nos (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 2 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 0
Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 — Skin And Appendages
Fungal Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Herpes Zoster (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin Carcinoma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 — Special Senses
Acute Kidney Failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 — Urogenital System
Genital Edema (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Kidney Function Abnormal (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Temsirolimus 175/75 mg (N=57) | Temsirolimus 175/25 mg (N=56) | Investigator's Choice (N=54) | Temsirolimus 175/25 mg Then 75 mg (N=3) | Investigator's Choice Then Temsirolimus 175/75 mg (N=4)
Abdominal Pain (General disorders) | 14 | 16 | 9 | 0 | 2 — Body As A Whole
Accidental Injury (General disorders) | 4 | 6 | 1 | 0 | 0
Asthenia (General disorders) | 38 | 34 | 13 | 3 | 1
Back Pain (General disorders) | 8 | 8 | 2 | 0 | 1
Cellulitis (General disorders) | 1 | 2 | 2 | 0 | 1
Chest Pain (General disorders) | 6 | 4 | 2 | 0 | 0
Chills (General disorders) | 14 | 5 | 6 | 0 | 0
Face Edema (General disorders) | 4 | 1 | 0 | 0 | 0
Fever (General disorders) | 21 | 16 | 17 | 0 | 2
Flu Syndrome (General disorders) | 2 | 5 | 1 | 0 | 0
Headache (General disorders) | 9 | 13 | 5 | 0 | 2
Hernia (General disorders) | 0 | 0 | 0 | 0 | 1
Infection (General disorders) | 17 | 15 | 3 | 0 | 2
Neoplasm (General disorders) | 2 | 3 | 0 | 0 | 0
Non-Specified Drug Reaction (General disorders) | 3 | 1 | 0 | 0 | 0
Pain (General disorders) | 19 | 13 | 2 | 1 | 2
Pelvic Pain (General disorders) | 0 | 3 | 1 | 0 | 0
Hemorrhage (Cardiac disorders) | 3 | 2 | 0 | 0 | 1 — Cardiovascular System
Hypertension (Cardiac disorders) | 2 | 5 | 0 | 0 | 0
Hypotension (Cardiac disorders) | 2 | 4 | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 5 | 4 | 2 | 0 | 0
Tachycardia Sinus (Cardiac disorders) | 1 | 3 | 0 | 0 | 0
Thrombophlebitis (Cardiac disorders) | 0 | 3 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 — Digestive System
Anorexia (Gastrointestinal disorders) | 23 | 17 | 8 | 1 | 0
Aphthous Stomatitis (Gastrointestinal disorders) | 3 | 4 | 0 | 0 | 0
Blood In Stool (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 9 | 4 | 10 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 26 | 19 | 6 | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 4 | 2 | 1 | 0 | 1
Dyspspsia (Gastrointestinal disorders) | 2 | 2 | 3 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 6 | 3 | 0 | 0 | 0
Melena (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 0
Mouth Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 3 | 5 | 0 | 0 | 0
Mucositis (Gastrointestinal disorders) | 21 | 9 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 14 | 17 | 11 | 1 | 2
Rectal Hemorrhage (Gastrointestinal disorders) | 5 | 1 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 12 | 6 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 8 | 7 | 3 | 0 | 2
Anemia (Blood and lymphatic system disorders) | 31 | 30 | 24 | 1 | 3 — Hemic And Lymphatic System
Ecchymosis (Blood and lymphatic system disorders) | 4 | 4 | 2 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 3 | 3 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 10 | 12 | 22 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 2 | 2 | 0 | 0
Lymphedema (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 3 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 7 | 7 | 10 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 15 | 19 | 22 | 2 | 1
Prothrombin Time Prolonged (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 45 | 47 | 29 | 3 | 4
Creatinine Increased (Metabolism and nutrition disorders) | 5 | 7 | 0 | 0 | 0 — Metabolic And Nutritional
Dehydration (Metabolism and nutrition disorders) | 2 | 4 | 0 | 0 | 0
Edema (Metabolism and nutrition disorders) | 3 | 6 | 6 | 0 | 0
Gamma Globulin Decreased (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0
Hypercholesteremia (Metabolism and nutrition disorders) | 11 | 10 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 6 | 6 | 0 | 1
Hyperlipemia (Metabolism and nutrition disorders) | 7 | 11 | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 5 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 14 | 10 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 7 | 6 | 0 | 0 | 0
Hypoproteinemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0 | 0
Lactic Dehydrogenase Increased (Metabolism and nutrition disorders) | 6 | 5 | 1 | 0 | 0
Peripheral Edema (Metabolism and nutrition disorders) | 14 | 13 | 9 | 0 | 1
SGOT Increased (Metabolism and nutrition disorders) | 2 | 6 | 1 | 0 | 0
SGPT Increased (Metabolism and nutrition disorders) | 1 | 3 | 1 | 0 | 0
Weight Gain (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Weight Loss (Metabolism and nutrition disorders) | 10 | 12 | 5 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 5 | 1 | 0 | 0 — Musculoskeletal System
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 1 | 1
Joint Disorder (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | 0
Leg Cramps (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 0 | 0
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 7 | 2 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 1 | 0 | 0
Anxiety (Nervous system disorders) | 9 | 4 | 3 | 0 | 0 — Nervous System
Depression (Nervous system disorders) | 5 | 5 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 6 | 1 | 0 | 0
Insomnia (Nervous system disorders) | 12 | 6 | 4 | 0 | 0
Neuropathy (Nervous system disorders) | 2 | 4 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 4 | 6 | 3 | 1 | 0
Sleep Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3 | 0 | 0 — Respiratory System
Cough Increased (Respiratory, thoracic and mediastinal disorders) | 19 | 18 | 5 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 | 12 | 16 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 26 | 16 | 3 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 7 | 9 | 4 | 0 | 0
Pleural Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 4 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 | 8 | 5 | 0 | 1
Pulmonary Physical Finding (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 2 | 0 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 3 | 0 | 0
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 0 | 0 | 0
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 2 | 0 | 2
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 5 | 2 | 0 | 0 | 0 — Skin And Appendages
Dry Skin (Skin and subcutaneous tissue disorders) | 7 | 5 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 6 | 1 | 2 | 1 | 0
Fungal Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 1 | 0
Herpes Simplex (Skin and subcutaneous tissue disorders) | 6 | 10 | 4 | 0 | 1
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 0 | 0
Nail Disorder (Skin and subcutaneous tissue disorders) | 11 | 10 | 1 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 5 | 3 | 4 | 0 | 0
Pruritic Rash (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 12 | 3 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 21 | 19 | 6 | 0 | 0
Skin Carcinoma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Skin Disorder (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 0 | 0
Sweating (Skin and subcutaneous tissue disorders) | 1 | 3 | 7 | 0 | 0
Abnormal Vision (Eye disorders) | 3 | 0 | 0 | 0 | 0 — Special Senses
Conjunctivitis (Eye disorders) | 4 | 2 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye Disorder (Eye disorders) | 3 | 0 | 0 | 0 | 0
Eye Hemorrhage (Eye disorders) | 3 | 1 | 0 | 0 | 0
Parosmia (Eye disorders) | 3 | 0 | 1 | 0 | 0
Taste Loss (Eye disorders) | 5 | 3 | 0 | 1 | 0
Taste Perversion (Eye disorders) | 9 | 2 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 4 | 5 | 1 | 0 | 0 — Urogenital System
Hematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 1
Urinary Frequency (Renal and urinary disorders) | 4 | 1 | 0 | 0 | 0
Urinary Tract Infection (Renal and urinary disorders) | 3 | 5 | 0 | 0 | 0
Local Reaction To Procedure (Investigations) | 3 | 3 | 1 | 1 | 0 — Adverse Event Associated with Miscellaneous factors

LIMITATIONS AND CAVEATS:
After the primary analysis was completed, efficacy data was no longer collected nor analyzed; Participants were followed for safety up to 6 months after the last dose of temsirolimus.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.